CLINICAL TRIAL: NCT02226380
Title: A Phase II Study of Neoadjuvant Chemotherapy With Modified FOLFOX6 Regimen and Effects of Tumor Regression in Locally Advanced Gastric Cancer
Brief Title: FOLFOX6 as Neoadjuvant Chemotherapy in Local Advanced Gastric Cancer
Acronym: FOLFOX6
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-JZ
Record Dates: First submitted 2014-08-24; First posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Gastric Cancer; Effects of Chemotherapy; Surgery
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mFOLFOX6,chemotherapy regimen (Experimental): oxaliplatin 85 mg/m2 and folinic acid 400 mg/m2 are administered intravenously for 2 hours on day 1 following by 5-FU at 2,400 mg/m2 by continuous infusion for 46hours every 2 weeks for 3 cycles before performing surgery
  Interventions: Drug: mFOLFOX6 regimen

INTERVENTIONS:
Drug: mFOLFOX6 regimen — oxaliplatin 85 mg/m2 and folinic acid 400 mg/m2 are administered intravenously for 2 hours on day 1 following by 5-FU at 2,400 mg/m2 by continuous infusion for 46hours every 2 weeks for 3 cycles before performing surgery

SUMMARY:
Purpose: This aim of the study is to evaluate the efficacy and safety of neoadjuvant chemotherapy with the modified FOLFOX6(mFOLFOX6) regimen and its impact on survival on a series in local advanced gastric cancer patients.

Patients and methods: The study is a prospective non-randomized study. Patients with histopathologically confirmed and locally advanced gastric cancer(T2-T4 or N+) are enrolled in the study. Patients are given mFOLFOX6 scheme for 3 cycles.A radical gastrectomy and a D2 lymphadenectomy was will be scheduled 3-6 weeks after the completion of the preoperative chemotherapy. Down-staging is assessed comparing pretreatment clinical staging with postoperative pathologic staging on patients who underwent radical surgery. Tumor down-staging and the grade of pathologic response are included in a statistical correlation between tumor regression induced by mFOLFOX6 neoadjuvant chemotherapy and survival.The primary endpoint is 3-year overall survival, secondary endpoints are disease-free survival, R0 resection rate, toxicity and prediction of response.

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria included histologically confirmed gastric cancer, the gastro-oesophageal junction(GEJ) may be involved, but the bulk of the tumour has to be in the stomach; age ≥18 years old, ECOG performance status score ≤2, no prior chemotherapy, TNM stage of T2-T4 or positive regional lymph nodes by endoscopic ultrasound or computed tomography (CT), and adequate hematological, heart, liver and renal functions (ALT and AST≤2.5 UNL, total bilirubin ≤1.5 UNL, and serum creatinine ≤1.5 UNL).

Exclusion Criteria:

Patients with second malignancies or evidence of severe or uncontrolled systemic disease were excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The 3-year overall survival rate in patients who will receive mFOLFOX6 regimen as neoadjuvant chemotherapy regimen | 3 years

SECONDARY OUTCOMES:
The 3-year disease-free survival rate in the patients who will receive mFOLFOX6 regimen neoadjuvant chemotherapy regimen | 3 year

OTHER OUTCOMES:
The R0 resection rate in the patients who will receive mFOLFOX6 regimen as neoadjuvant chemotherapy regimen | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Wang, Master, Study Director — Department of Medical Oncology Peking Union Medical College Hospital
Locations (2):
- China (2):
  - Department of Oncology and Surgery, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality

REFERENCES:
- [Result] Li ZY, Koh CE, Bu ZD, Wu AW, Zhang LH, Wu XJ, Wu Q, Zong XL, Ren H, Tang L, Zhang XP, Li JY, Hu Y, Shen L, Ji JF. Neoadjuvant chemotherapy with FOLFOX: improved outcomes in Chinese patients with locally advanced gastric cancer. J Surg Oncol. 2012 Jun 15;105(8):793-9. doi: 10.1002/jso.23009. Epub 2011 Dec 20. PMID 22189752